CLINICAL TRIAL: NCT02088021
Title: Assessment of the St. Jude Medical PorticoTM Re-sheathable Aortic Valve System - Alternative Access
Acronym: PorticoALTEU
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL07045
Record Dates: First submitted 2014-03-04; First posted 2014-03-14 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Symptomatic Aortic Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Portico Transcatheter Aortic Valve Implantation (Experimental): Placement of the SJM Portico aortic valve with a ALC delivery system
  Interventions: Device: Portico Transcatheter Aortic Valve

INTERVENTIONS:
Device: Portico Transcatheter Aortic Valve — Placement of the SJM Portico aortic valve with a ALC delivery system

SUMMARY:
The purpose of this clinical investigation is to evaluate the use of the Portico ALC Delivery System to place a transcatheter aortic valve through an alternative access site, specifically subclavian/axillary or TAo.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent.
* Subject is 65 years of age or older at the time of index procedure, and/or has comorbidities that, in the opinion of the Principal Investigator or the Subject Selection Committee, preclude surgical valve replacement.
* Subject's aortic annulus diameter meets the range indicated in the Instructions for Use as measured by multislice CT conducted within 120 days prior to the index procedure.
* Subject has senile degenerative aortic stenosis with echocardiography within 30 days of index procedure as defined by at least 1 of the following:

  * derived mean gradient greater than 40 mmHg, OR
  * jet velocity greater than 4.0 m/s, OR
  * aortic valve area of less than 0.8 cm2, OR
  * aortic valve area index less than or equal to 0.6 cm2/m2.
* Subject has symptomatic aortic stenosis as demonstrated by NYHA Functional Classification of II, III, or IV.
* Subject is deemed high operable risk and delivery route is suitable for TAVI per the medical opinion of the Subject Selection Committee.
* Subject's predicted operative mortality or serious, irreversible morbidity risk is less than 50% at 30 days post index procedure.

Exclusion Criteria:

* Subject is unwilling or unable to comply with all study-required follow-up evaluations.
* Subject has a documented history of a cerebral vascular accident (CVA) or transient ischemic attack (TIA) within 6 months (less than or equal to 180 days) prior to the index procedure.
* Subject has carotid artery disease requiring intervention.
* Evidence of an acute myocardial infarction (MI) within 30 days prior to patient providing consent (defined as: ST Segment Elevation as evidenced on 12 Lead ECG).
* Subject has a native aortic valve that is congenitally unicuspid, bicuspid, quadricuspid or non-calcified as seen by echocardiography.
* Subject has mitral valvular regurgitation greater than grade III.
* Subject has moderate or severe mitral stenosis.
* Subject has a pre-existing prosthetic cardiac device, valve, or prosthetic ring in any position.
* Subject refuses any blood product transfusion.
* Subject refuses surgical valve replacement.
* Subject has left ventricular ejection fraction (LVEF) less than 20%.
* Subject has documented, untreated symptomatic coronary artery disease (CAD) requiring revascularization.
* Subject has had a percutaneous interventional or other invasive cardiovascular or peripheral vascular procedure less than or equal to 14 days of index procedure.
* Subject has severe basal septal hypertrophy that would interfere with transcatheter aortic valve placement.
* Subject has a history of, or is currently diagnosed with endocarditis.
* There is imaging evidence of intracardiac mass, thrombus, or vegetation.
* Subject is considered hemodynamically unstable (requiring inotropic support or mechanical heart assistance).
* Subject is in acute pulmonary edema or requiring intravenous diuretic therapy to stabilize heart failure.
* Subject with significant pulmonary disease as determined and documented by the Investigator.
* Subject has significant chronic steroid use as determined and documented by the Investigator.
* Subject has a documented hypersensitivity or contraindication to anticoagulant or antiplatelet medication.
* Subject has renal insufficiency as evidenced by a serum creatinine greater than 3.0 mg/dL (265.5 µmol/L) or end-stage renal disease requiring chronic dialysis.
* Subject has morbid obesity defined as a BMI greater than or equal to 40.
* Subject has ongoing infection or sepsis.
* Subject has blood dyscrasias (eg, leukopenia, acute anemia, thrombocytopenia, history of bleeding diathesis, or coagulopathy).
* Subject has a current autoimmune disease that, in the opinion of the Principal Investigator or the Subject Selection Committee, precludes the subject from study participation.
* Significant ascending aortic disease documented by diameter greater than 40mm.
* Subject has an active peptic ulcer or has had gastrointestinal (GI) bleeding within 90 days prior to the index procedure.
* Subject is currently participating in another investigational drug or device study.
* Subject requires emergency surgery for any reason.
* Subject has a life expectancy less than 12 months.
* Subject has other medical, social or psychological conditions that, in the opinion of the Principal Investigator or the Subject Selection Committee, preclude the subject from study participation.
* Subject is diagnosed with dementia or admitted to a chronic care facility which would fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits.
* Subject is unwilling or unable to comply with all study-required follow-up evaluations.
* Subject has a documented history of a cerebral vascular accident (CVA) or transient ischemic attack (TIA) within 6 months (less than or equal to 180 days) prior to the index procedure.
* Subject has carotid artery disease requiring intervention.
* Evidence of an acute myocardial infarction (MI) within 30 days prior to patient providing consent (defined as: ST Segment Elevation as evidenced on 12 Lead ECG).
* Subject has a native aortic valve that is congenitally unicuspid, bicuspid, quadricuspid or non-calcified as seen by echocardiography.
* Subject has mitral valvular regurgitation greater than grade III.
* Subject has moderate or severe mitral stenosis.
* Subject has a pre-existing prosthetic cardiac device, valve, or prosthetic ring in any position.
* Subject refuses any blood product transfusion.
* Subject refuses surgical valve replacement.
* Subject has left ventricular ejection fraction (LVEF) less than 20%.
* Subject has documented, untreated symptomatic coronary artery disease (CAD) requiring revascularization.
* Cardiovascular or peripheral vascular procedure less than or equal to 14 days of index procedure.
* Subject has severe basal septal hypertrophy that would interfere with transcatheter aortic valve placement.
* Subject has a history of, or is currently diagnosed with endocarditis.
* There is imaging evidence of intracardiac mass, thrombus, or vegetation.
* Subject is considered hemodynamically unstable (requiring inotropic support or mechanical heart assistance).
* Subject is in acute pulmonary edema or requiring intravenous diuretic therapy to stabilize heart failure.
* Subject with significant pulmonary disease as determined and documented by the Investigator.
* Subject has significant chronic steroid use as determined and documented by the Investigator.
* Subject has a documented hypersensitivity or contraindication to anticoagulant or antiplatelet medication.
* Subject has renal insufficiency as evidenced by a serum creatinine greater than 3.0 mg/dL (265.5 µmol/L) or end-stage renal disease requiring chronic dialysis.
* Subject has morbid obesity defined as a BMI greater than or equal to 40.
* Subject has ongoing infection or sepsis.
* Subject has blood dyscrasias (eg, leukopenia, acute anemia, thrombocytopenia, history of bleeding diathesis, or coagulopathy).
* Significant ascending aortic disease documented by diameter greater than 40mm.
* Subject has an active peptic ulcer or has had gastrointestinal (GI) bleeding within 90 days prior to the index procedure.
* Subject is currently participating in another investigational drug or device study.
* Subject requires emergency surgery for any reason.
* Subject has a life expectancy less than 12 months.
* Subject has other medical, social or psychological conditions that, in the opinion of the Principal Investigator or the Subject Selection Committee, preclude the subject from study participation.
* Subject is diagnosed with dementia or admitted to a chronic care facility which would fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits.
* Subject has a documented allergy to contrast media, nitinol alloys, porcine tissue, or bovine tissue.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Major Vascular Complications related to the Portico ALC Delivery System | 30 day post procedure
All cause mortality | 30 day post procedure

SECONDARY OUTCOMES:
Event Rates | 30 days post procedure
  Event rates as described by VARC-2
  "Updated standardized endpoint definitions for transcatheter aortic valve implantation: the Valve Academic Research Consortium-2 consensus document European Heart Journal (2012) 33, 2403-2418."
Functional improvement from baseline | 30 days post procedure
  Functional improvement from baseline as compared to 30 days by:
  * NYHA Functional Classification
  * Six Minute Walk Test
  * Effective Orifice Area (EOA)
Acute device success | 12 months post procedure
  Acute device success defined as:
  * Ability of the Portico ALC Delivery System to successfully deliver, deploy, and resheath (if necessary) a transcatheter aortic valve
  * Absence of procedural mortality
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location
  * Intended performance of the prosthetic heart valve, as defined by:
  * mean aortic valve gradient <20 mmHg or peak velocity <3 m/s, and
  * no moderate or severe prosthetic valve regurgitation

CONTACTS AND LOCATIONS:
Overall Officials: Axel Linke, Prof Dr. med, Principal Investigator — Heart Center Leipzig - University Hospital